CLINICAL TRIAL: NCT02084914
Title: The Effect of Endometrial Scratching by Pipelle on Pregnancy Rate in Couples With Unexplained Infertility
Brief Title: Endometrial Scratching by Pipelle on Pregnancy Rate in Unexplained Infertility
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Elsayed Hassan Elbohoty, Lecturer in OB GYN, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ESBPOPRIUI
Record Dates: First submitted 2014-03-10; First posted 2014-03-12 (Estimated); Last update posted 2014-03-12 (Estimated); Status verified 2014-03

CONDITIONS: Unexplained Infertility
Keywords: endometrial scratching; pipelle; pregnancy rate; unexplained infertility

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental): Endometrial scraching of uterine cavity by pipelle .
  Interventions: Procedure: Endometrial scratching
- Group B (Active Comparator): Uterine sound intoduced into uterine cavity without scratch .
  Interventions: Procedure: Endometrial scratching

INTERVENTIONS:
Procedure: Endometrial scratching — Group A: pipelle Group B: sound
  Other Names: Unexplained Infertility

SUMMARY:
Research question:

Population: women with unexplained infertility. Intervention: endometrial scratching by pipelle for women with unexplained infertility.

Comparison: to compare with non endometrial scratching for women with unexplained infertility.

Outcome: the biochemical pregnancy rate.

Research hypothesis:

Null hypothesis: there is no difference in the rate of pregnancy between scratching and non endometrial scratching in women with unexplained infertility.

Alternative hypothesis: there is difference in the rate of pregnancy between scratching and non endometrial scratching in women with unexplained infertility.

DETAILED DESCRIPTION:
Unexplained infertility (UI) is a term used to describe infertile couples in whom standard investigations, including semen analysis, tests of ovulation and tubal patency, have failed to detect any gross abnormality (Crosignani et al., 1993). It is a diagnosis of exclusion, almost 30-40% of infertile couples would suffer from this type of subfertility (Simth et al., 2003). A diversity of causes had been hypothesized to explain the condition. Cervical, uterine, ovulatory, peritoneal, immunological, endocrinological, genetic defects and reproductive physiology disturbances had been continuously suggested as potential causative factors (Rov et al., 2005; Shveiky et al., 2006; Bellver et al., 2008; Golubovsky, 2008; Woodson, 2008). Empirically, interventions for managing unexplained infertility had been widely practiced. These interventions include expectant management, intrauterine insemination (IUI) with ovarian stimulation and in vitro fertilization (El-Toukhy & Khalaf, 2008; Bhattachary et al., 2010).

In humans, the uterus becomes receptive during the midsecretory phase of the menstrual cycle (days 19-23), commonly known as the window of implantation (WOI). It is assumed that inadequate uterine receptivity is responsible for approximately two-thirds of implantation failures (Simon et al., 1998). Since an impairment of endometrial receptivity may be a cause of subfertility in a group of couples diagnosed with unexplained infertility (Jasper et al., 2006; Boroujerdnia & Nikbakht, 2008; Konac et al., 2009). Endometrial scratching may help a group of couples with unexplained infertility.

ELIGIBILITY:
Inclusion Criteria 1. Women diagnosed to have unexplained infertility aged between 20-35y.

2. Regular menstruation with the length of the cycle between 21-35 days. 3. Ovulation confirmed by appropriately timed mid-luteal progesterone. 4. Fertile semen variables (according to world health organization criteria 2010).

5. Bilateral tubal patency (demonstrated by laparoscopy or hystrosalpingography).

Exclusion Criteria: 1- Patients aged less than 20 y. or more than 35y 2- Infertile semen analysis. 3- Abnormal hormonal profile (FSH level more than 10). 4- Patient diagnosed as polycystic ovary (PCO). 5- Medical disorders as hypertention,liver and renal diseases. 6- Endocrinal disorders as hyperthyroidism,hypothyroidism and diabetes mellitus.

7- Pelvic pathology as PID or uterine fibroids. 8- No previous history or planning for IVF. 9- Unwilling to comply with the protocol. 10- Participation in another clinical trial in the last 3 months prior to the start of this study.

-

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 158 (Estimated)
Dates: Start 2013-12; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Biochemical Pregnancy Rate in Scratching and Non Endometrial Scratching Group. | six months

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed E Elbohoty, MD, Principal Investigator — OB GYN Department, faculty of Medicine, ASU
Locations (1):
- Ain Shams Maternity Hospital, Cairo, Egypt